CLINICAL TRIAL: NCT06669728
Title: Diagnostic Efficacy of Deep Neural Network Algorithm Based on Preoperative Scheimpflug-based Anterior Segment Image for Implantable Collamer Lens Selection and Prediction
Brief Title: Study on the Diagnostic Efficacy of ICL Selection and Prediction Depth Model Based on Eye Images
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Jian Xiong, Associate research fellow; Attending physician, Second Affiliated Hospital of Nanchang University
Other Study IDs: [2024] NO.(93)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-01

CONDITIONS: Posterior Chamber Phakic Intraocular Lens; Vault; Deep Neural Network; Myopia; Anterior Chamber Angle
Keywords: Posterior Chamber Phakic Intraocular Lens; Vault; Deep Neural Network
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eyes with ICL surgeries: Eyes with SMILE surgeries which were performed by surgeons with experiences.
  Interventions: Diagnostic Test: AI diagnostic algorithm

INTERVENTIONS:
Diagnostic Test: AI diagnostic algorithm — The ICL procedures collected would be assessed by the algorithm. The performance of the algorithm would be assessed, including accuracy, AUC, sensitivity and specificity.

SUMMARY:
To evaluate the diagnostic efficacy of deep learning network model in implantable collamer lens selection and prediction in a multicenter cross-sectional study

DETAILED DESCRIPTION:
Posterior chamber intraocular lens implantation is an main choice for myopia correction. Implantable collamer lens (ICL) is currently the most widely used, and the official reference index is mainly based on biological parameters obtained from eye images. The parameter acquisition and selection of ICL design are often controversial, forcing the doctors to synthesize multiple modal data, making the optimization of ICL formula being a focus of attention in refractive surgery. This research aimed to build an image-based ICL prediction algorithm to assist human physicians in decision-making and improve the accuracy, safety and predictability of ICL implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years ;
2. Myopia, with or without astigmatism, annual diopter change ≤ 0.50 D for 2 consecutive years ;
3. Anterior chamber depth ≥ 2.80 mm ;
4. Corneal endothelial cell count ≥ 2000 / mm2, stable cell morphology ;
5. There were no other ocular diseases that significantly affected vision and / or systemic organic lesions that affected surgical recovery.

Exclusion Criteria:

1. There were no other ocular diseases that significantly affected vision and / or systemic organic lesions that affected surgical recovery;
2. Have a history of corneal refractive surgery or intraocular surgery ;
3. Corneal endothelial cell count is low ;
4. Those with systemic diseases ;
5. Lactating or pregnant women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from clinics in different eye centers across China. Each subject must with complete surgical video recording and medical records.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
AUROC of convolutional neural network in predicting vault after ICL surgery | Day 7
  The area under the receiver operating characteristic of convolutional neural network in predicting vault after ICL surgery
AUROC of convolutional neural network in predicting anterior chamber angle after ICL implantation | Day 7
  The area under the receiver operating characteristic of convolutional neural network in predicting anterior chamber angle after ICL implantation

SECONDARY OUTCOMES:
Sensitivity and specificity of convolutional neural network in predicting Vault after ICL implantation | Day 7
  Sensitivity and specificity of convolutional neural network in predicting Vault after ICL implantation
Sensitivity and specificity of convolutional neural network in predicting anterior chamber angle after ICL implantation | Day 7
  Sensitivity and specificity of convolutional neural network in predicting anterior chamber angle after ICL implantation

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No